CLINICAL TRIAL: NCT03857854
Title: A Phase III, Randomized, Double-blind, Placebo Controlled, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Pirfenidone in Subjects With Dermatomyositis Interstitial Lung Disease (Dm-ILD)
Brief Title: Efficacy and Safety of Pirfenidone in Patient With Dermatomyositis Interstitial Lung Disease (Dm-ILD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNI-F647-1702
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Dermatomyositis Interstitial Lung Disease (Dm-ILD)
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): pirfenidone group
  Interventions: Drug: Pirfenidone
- placebo group (Placebo Comparator): control group
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Pirfenidone — treatment group
  Arms: treatment group
Drug: Placebos — placebo group
  Arms: placebo group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pirfenidone in subjects with dermatomyositis interstitial lung disease

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects aged between 18 and 65 years of age
2. According to the 1975 Borhan and Peter inflammatory myopathy diagnosed as dermatomyositis classification criteria (dermatomyositis, DM); or according to the revised clinical criteria for diagnosis of Sontheimer disease dermatomyositis (CADM).
3. The diagnosis of pulmonary related Interstitial Lung Disease confirmed by HRCT
4. Forced vital capacity (FVC) 40% to 80% predicted(include 40% and80% )
5. Carbon monoxide diffusing capacity (DLco) 30% to 89% of predicted normal(include 30% and89% )
6. Has received Glucocorticoid (hereinafter referred to as the "hormone") and at least one immunosuppressive therapy for more than 3 months, the hormone dosage (prednisone equivalent dose calculation) should be less than 15mg/d for at least 1 months, should be immunosuppressant cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine and at least one of methotrexate in, and the type and dose of immunosuppressive agents should be at least stable more than 3 months. The hormone and immunosuppressant therapy scheme allows a reduction in the study period, but is not allowed to increase the volume.
7. Women of childbearing age must agree and promise to use the form of medical care for at least 3 months after the trial, during the entire study period (including follow-up), and at the end of the trial.
8. Patients volunteered to participate in the trial, with good compliance and ability to understand and sign informed consent before the study.

Exclusion Criteria:

1. Subjects not fulfill all of the above inclusion criteria
2. Combined with other rheumatic diseases such as systemic sclerosis, systemic lupus erythematosus, Sjogren's syndrome, mixed connective tissue disease, undifferentiated connective tissue disease, and systemic vasculitis, such as ANCA associated vasculitis.
3. Combined with other muscle diseases and may cause symptoms of myasthenia gravis disease, including neurological diseases (such as muscular dystrophy, myasthenia gravis, amyotrophic lateral sclerosis, Guillain Barre syndrome), cancer, drugs (such as statins), infection, genetic diseases, endocrine disorders, electrolyte disorder rhabdomyolysis.
4. The clinical history, signs, serological examination, HRCT and bronchoalveolar lavage results suggest that in addition to inflammatory myopathy and other diseases caused by ILD, such as CTD, systemic vasculitis, infection, tumor, allergic pneumonia caused by sarcoidosis or environmental factors.
5. Combined viscera function significantly abnormal patient:

   1. Liver:AST, ALT >1.3ULN;Bilirubin >1.5 ULN; Cirrhosis of the liver class for Child Pugh C;
   2. Kidney:Creatinine clearance <30 mL/min;
   3. Lung:Airway obstruction (pre-bronchodilator FEV1/FVC <0.7);Other clinically significant pulmonary abnormalities;
   4. Cardiovascular:i.Six weeks in severe hypertension, and out of control after treatment(≥160/100mmHg);ii.Myocardial infarction within six months;iii.A period of 6 Months in unstable angina;iv.pulmonary artery hypertension and right heart failure were significant;
   5. Gastrointestinal tract: with active peptic ulcer;
   6. Nervous system: Patients with psychiatric disorders;
   7. The blood coagulation function: History of thrombotic event within last year(Including stroke and transient ischemic attack).
6. Researchers, for other diseases (not inflammatory myopathy, such as malignant tumor) and make the life expectancy of < 1 year of patients
7. Allergic to test drugs or components (e.g. lactose)
8. Patients with actinic dermatitis
9. Previous treatment with nintedanib or pirfenidone
10. Within 3 months to participate in other clinical trials;
11. Combined medication: hormone > 15mg/d, were less than 1 months before a stable dose of patients; the use of other immunosuppressive agents (except cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, methotrexate and) patients; immunosuppression stable < 3 months; during the study of hormones and immunosuppressive agents are likely to increase patients.
12. Major surgery is planned during the treatment period.
13. Pregnancy or lactation or make a schedule during the trials.
14. Give the drug 28 days before or after administration of the 3 month period, women of childbearing age * are unwilling or unable to use contraceptive methods highly effective (according to ICH M3 (R2)), a highly effective means in the correct and consistent application of a barrier method when the failure rate of less than 1% per year. * women of childbearing age is defined has undergone menarche and in line with "infertile women" standard "[female infertile women" is defined as: postmenopausal period (12 months without menstruation, no other medical reasons) or permanent sterilization (e.g., tubal occlusion, hysterectomy, bilateral ovarian resection or bilateral tubal resection women)].
15. According to the researchers,exhibited evidence of alcohol or drug abuse.
16. Patients who were unable to understand or comply with the study procedures, including the completion of a self-administered questionnaire in the absence of help, were less likely to complete the trial.
17. Severe limb weakness or joint disease that affects the stability and endurance of a patient who is unable to perform a 6 minute walking test.
18. Clinical signs of malabsorption or needing parenteral nutrition.
19. Patients who were unable to cope with pulmonary function tests.
20. With mental illness .
21. Researchers determined that they did not participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Relative change from baseline (%) of FVC | 52 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang, Ling, Beijing, Beijing Municipality, China